CLINICAL TRIAL: NCT02819271
Title: A First-in-Human Study of the Safety of Single Continuous Intravenous Infusions of CXL-1427 for up to 48 Hours in Healthy Volunteers
Brief Title: A First-in-Human Study of the Safety of Single Continuous Intravenous (IV) Infusions of CXL-1427 for up to 48 Hours in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Cardioxyl Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXL-1427-01; CV013-005 (Other: BMS)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXL-1427 (BMS-986231) (Experimental): Experimental
  Interventions: Drug: CXL-1427 Ascending Dose; Drug: CXL-1427 Descending Dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CXL-1427 Ascending Dose
  Other Names: BMS-986231
  Arms: CXL-1427 (BMS-986231)
Other: Placebo
  Arms: Placebo
Drug: CXL-1427 Descending Dose
  Other Names: BMS-986231
  Arms: CXL-1427 (BMS-986231)

SUMMARY:
This study is designed to assess a safe dosage of the drug CXL-1427 (BMS-986231) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of any acute or chronic health disorder
* Not have taken any prescription medication within 15 days of study entry
* Not have taken any over-the-counter medication or herbal/vitamin supplement within 3 days of study entry
* Not have not have any dietary restrictions
* Have a body mass index (BMI) of ≥18 to ≤34
* Weigh at least 50kg (110 pounds)

Exclusion Criteria:

* Be a current or recent (within 6 months of the Screening Visit) smoker or user of any nicotine-containing product
* Have a history of symptomatic hypotension, orthostatic hypotension or syncope
* Have a history of headaches or other symptoms attributable to caffeine withdrawal
* Have a history of any bleeding diathesis
* Have a positive serology screen for HIV antibody, hepatitis B surface antigen or hepatitis C antibody at screening

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety measured by percentage of Treatment Emergent Adverse Events (TEAEs) | Up to 31 days
Tolerability measured by percentage of Treatment Emergent Adverse Events (TEAEs) | Up to 31 days

SECONDARY OUTCOMES:
Steady-state plasma concentration (Css) | Up to 4 days
Area under the plasma concentration (AUC) vs. time curve | Up to 4 days
Terminal elimination half-life (1/2) | Up to 4 days
Total body clearance (CL) | Up to 4 days
Steady-state volume of distributions (Vss) | Up to 4 days
Time to Css | Up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Cardioxyl Pharmaceuticals, Study Director — Cardioxyl Pharmaceuticals